CLINICAL TRIAL: NCT00776009
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled, Cross-over Study Evaluating the Safety and Efficacy of Dex-Methylphenidate Extended Release 30 mg vs. 20 mg as Measured by SKAMP-Combined Scores in Children With Attention-Deficit/Hyperactivity Disorder (ADHD) in a Laboratory Classroom Setting.
Brief Title: Efficacy and Safety of Dex-Methylphenidate Extended Release 30 mg Versus 20 mg in Children (6-12 Years) With Attention-Deficit/Hyperactivity Disorder (ADHD) in a Laboratory Classroom Setting.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Study Director Novartis Pharmaceuticals, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRIT124EUS21
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD, children, subjects, laboratory classroom
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Dex-Methylphenidate hydrochloride (Focalin® XR) 30 mg (Experimental): Dex-Methylphenidate hydrochloride (Focalin® XR) 30 mg dose (one 20 mg capsule and one 10 mg capsule) orally once a day for 7 days.
  Interventions: Drug: Dex-Methylphenidate hydrochloride Extended Release (Focalin® XR)
- Dex-Methylphenidate hydrochloride (Focalin® XR) 20 mg (Active Comparator): Dex-Methylphenidate hydrochloride (Focalin® XR) one 20 mg capsule orally once a day for 7 days.
  Interventions: Drug: Dex-Methylphenidate hydrochloride Extended Release (Focalin® XR)
- Placebo (Placebo Comparator): Two Capsules taken orally once a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dex-Methylphenidate hydrochloride Extended Release (Focalin® XR) — 10 mg and/or 20 mg capsules
  Arms: Dex-Methylphenidate hydrochloride (Focalin® XR) 20 mg; Dex-Methylphenidate hydrochloride (Focalin® XR) 30 mg
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of Dex-Methylphenidate Extended Release 30 mg compared to 20 mg in pediatric patients ages 6-12 with Attention-Deficit Hyperactivity Disorder (ADHD) in a 12-hour laboratory classroom setting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 6-12 years, inclusive.
* Subjects meeting the DSM-IV criteria for primary diagnosis of ADHD-Combined type, or predominantly hyperactive-impulsive subtype, as established by the K-SADS-PL (Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version). If a DSM-IV-defined ADHD diagnosis is difficult to establish due to possible co-morbidity, the subject will not be enrolled into the study.
* Subjects should be on a stabilized total daily dose or nearest equivalent of 40-60 mg methylphenidate or 20-30 mg of d-methylphenidate for at least two weeks prior to Screening visit.

Exclusion Criteria:

* Subject or subject's guardian unable to understand or follow instructions necessary to participate in the study.
* Diagnosed with or history of a tic disorder or Tourette's syndrome.
* History of seizure disorder.
* The presence of a known medical condition that would preclude the use of methylphenidate.
* A history (within the past year) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurological disease.
* ALT (Alanine Amino Transferase), AST (Aspartate Amino Transferase), GGT (Gamma glutamyl transferase) or serum creatinine greater then 2X the ULN (Upper Limit of Normal) at Screening.
* A history of psychiatric illness or substance use disorder (e.g., schizophrenia, bipolar disorder, autism, abuse or dependence, depression, severe Conduct Disorder or severe Oppositional defiant disorder)
* Subjects who have participated in an investigational trial within the past 4 weeks (28 days)
* Subjects who are currently taking antidepressants or other psychotropic medication.
* Subjects who have initiated psychotherapy during the three months prior to randomization.
* Subjects with a positive urine drug screen.
* Subjects who have a history of poor response or intolerance to methylphenidate or d-methylphenidate.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (8):
- United States (8):
  - Clinical Study Center, LLC, Little Rock, Arkansas
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Miami Research Associates, South Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Houston, Texas
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - Behavioral Neurology, Lubbock, Texas

REFERENCES:
- [Derived] Brams M, Turnbow J, Pestreich L, Giblin J, Childress A, McCague K, Muniz R. A randomized, double-blind study of 30 versus 20 mg dexmethylphenidate extended-release in children with attention-deficit/hyperactivity disorder: late-day symptom control. J Clin Psychopharmacol. 2012 Oct;32(5):637-44. doi: 10.1097/JCP.0b013e3182677825. PMID 22926597

RESULTS

PARTICIPANT FLOW:
Groups:
- Focalin XR 20 mg First, Then Focalin XR 30 mg, Then Placebo: Period 1: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days followed by Period 2: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days followed by Period 3: Placebo orally once a day for 7 days.
- Focalin XR 30 mg First, Then Placebo, Then Focalin XR 20 mg: Period 1: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days followed by Period 2: Placebo orally once a day for 7 days followed by Period 3: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days.
- Focalin XR 30 mg First, Then Focalin XR 20 mg, Then Placebo: Period 1: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days followed by Period 2: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days followed by Period 3: Placebo orally once a day for 7 days .
- Placebo First, Then Focalin XR 20 mg, Then Focalin XR 30 mg: Period 1: Placebo orally once a day for 7 days followed by Period 2: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days followed by Period 3: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days.
- Focalin XR 20 mg First, Then Placebo, Then Focalin XR 30 mg: Period 1: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days followed by Period 2: Placebo orally once a day for 7 days followed by Period 3: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days.
- Placebo First, Then Focalin XR 30 mg, Then Focalin XR 20 mg: Period 1: Placebo orally once a day for 7 days followed by Period 2: Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days followed by Period 3: Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days.
Period: Period 1: First Intervention
Arm/Group | Focalin XR 20 mg First, Then Focalin XR 30 mg, Then Placebo | Focalin XR 30 mg First, Then Placebo, Then Focalin XR 20 mg | Focalin XR 30 mg First, Then Focalin XR 20 mg, Then Placebo | Placebo First, Then Focalin XR 20 mg, Then Focalin XR 30 mg | Focalin XR 20 mg First, Then Placebo, Then Focalin XR 30 mg | Placebo First, Then Focalin XR 30 mg, Then Focalin XR 20 mg
Started | 26 | 28 | 29 | 27 | 28 | 27
Completed | 26 | 27 | 28 | 27 | 26 | 27
Not Completed | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1 | 0
Period: Period 2: Second Intervention
Arm/Group | Focalin XR 20 mg First, Then Focalin XR 30 mg, Then Placebo | Focalin XR 30 mg First, Then Placebo, Then Focalin XR 20 mg | Focalin XR 30 mg First, Then Focalin XR 20 mg, Then Placebo | Placebo First, Then Focalin XR 20 mg, Then Focalin XR 30 mg | Focalin XR 20 mg First, Then Placebo, Then Focalin XR 30 mg | Placebo First, Then Focalin XR 30 mg, Then Focalin XR 20 mg
Started | 26 | 27 | 28 | 27 | 26 | 27
Completed | 25 | 27 | 27 | 27 | 26 | 26
Not Completed | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0
Period: Period 3: Third Intervention
Arm/Group | Focalin XR 20 mg First, Then Focalin XR 30 mg, Then Placebo | Focalin XR 30 mg First, Then Placebo, Then Focalin XR 20 mg | Focalin XR 30 mg First, Then Focalin XR 20 mg, Then Placebo | Placebo First, Then Focalin XR 20 mg, Then Focalin XR 30 mg | Focalin XR 20 mg First, Then Placebo, Then Focalin XR 30 mg | Placebo First, Then Focalin XR 30 mg, Then Focalin XR 20 mg
Started | 25 | 27 | 27 | 27 | 26 | 26
Completed | 24 | 27 | 27 | 27 | 26 | 26
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Focalin XR 20 mg First, Then Focalin XR 30 mg, Then Placebo | Focalin XR 30 mg First, Then Placebo, Then Focalin XR 20 mg | Focalin XR 30 mg First, Then Focalin XR 20 mg, Then Placebo | Placebo First, Then Focalin XR 20 mg, Then Focalin XR 30 mg | Focalin XR 20 mg First, Then Placebo, Then Focalin XR 30 mg | Placebo First, Then Focalin XR 30 mg, Then Focalin XR 20 mg | Total
Number analyzed (Participants) | 26 | 28 | 29 | 27 | 28 | 27 | 165
Age Continuous [Mean (Standard Deviation); unit: Years] | 9.3 (1.7) | 9.4 (1.7) | 10.0 (1.8) | 9.4 (2.0) | 9.5 (1.8) | 9.6 (2.0) | 9.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 10 | 10 | 12 | 14 | 71
  Male | 17 | 12 | 19 | 17 | 16 | 13 | 94
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 29 | 27 | 28 | 27 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-dose in the Swanson, Kotkin, Agler, M Flynn, and Pelham (SKAMP) Combined Attention and Deportment Scores at 10, 11, and 12 Hour (Averaged) Post-dose
Description: SKAMP is a 13-item rating scale that measures classroom manifestations of ADHD consisting of 2 subscales (7 items for Attention and 6 items for Deportment) used to generate a score at Hours 10, 11 and 12 on Day 7 of Weeks 1, 2 and 3. The ratings were based on both frequency and quality of specific behaviors. The rating scale is 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 78. The reported measure is the difference from baseline of the 2 combined subscores averaged over Hours 10, 11 and 12. A negative score indicates improvement.
Time Frame: Pre-dose to 10, 11, and 12 hours post-dose
Population: Intent-to-treat population included all randomized patients who took at least 1 dose of study medication and who had at least 1 post-dose efficacy measurement
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg: Summary of the one week treatment on Dex-Methylphenidate hydrochloride (Focalin XR) 20 mg dose orally once a day for 7 days for all participants regardless of sequence.
- Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg: Summary of the one week treatment on Dex-Methylphenidate hydrochloride (Focalin XR) 30 mg dose orally once a day for 7 days for all participants regardless of sequence.
- Placebo: Summary of the one week treatment on Placebo orally once a day for 7 days for all participants regardless of sequence.
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Placebo
Number analyzed (Participants) | 159 | 158 | 158
Scores on a scale | -2.02 (0.717) | -4.47 (0.724) | 4.50 (.723)

2. Secondary Outcome: Change From Pre-dose in the Swanson, Kotkin, Agler, M Flynn, and Pelham (SKAMP) Attention Score at 10, 11, and 12 Hour (Averaged) Post-dose
Description: SKAMP is a 13-item rating scale consisting of 2 subscales (7-items for Attention and 6-items for Deportment) that measures classroom manifestations of ADHD. SKAMP was used to generate a score on the Attention subscale at Hours 10, 11, and 12 on Day 7 of Weeks 1, 2, and 3. The rating scale is 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 42 for the Attention subscale. The reported measure is the difference from baseline of the subscore averaged over Hours 10, 11, and 12. A negative score indicates improvement.
Time Frame: Pre-dose to 10, 11, and 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Placebo
Number analyzed (Participants) | 159 | 158 | 158
Scores on a scale | -1.33 (0.397) | -2.62 (0.400) | 0.94 (0.405)

3. Secondary Outcome: Change From Pre-dose in the Swanson, Kotkin, Agler, M Flynn, and Pelham (SKAMP) Deportment Score at 10, 11, and 12 Hour (Averaged) Post-dose
Description: SKAMP is a 13-item rating scale consisting of 2 subscales (7-items for Attention and 6-items for Deportment) that measures classroom manifestations of ADHD. SKAMP was used to generate a score on the Deportment subscale at Hours 10, 11, and 12 on Day 7 of Weeks 1, 2, and 3. The rating scale is 0 (normal, no impairment) to 6 (maximum impairment) for a total possible combined score of 0 to 36 for the Deportment subscale. The reported measure is the difference from baseline of the subscore averaged over Hours 10, 11, and 12. A negative score indicates improvement.
Time Frame: Pre-dose to 10, 11, and 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Placebo
Number analyzed (Participants) | 159 | 158 | 158
Scores on a scale | -0.39 (0.423) | -1.49 (0.426) | 2.95 (0.424)

4. Secondary Outcome: Change From Pre-dose in the Permanent Product Measure of Performance of Measurement (PERMP) Math Test-Attempted Score at 10, 11, and 12 Hours (Averaged) Post-dose
Description: Permanent Product Measure of Performance of Measurement (PERMP) is an age-adjusted, paper-and-pencil math test consisting of 5 pages of 80 math problems each presented in ascending order of difficulty (requiring addition, subtraction, multiplication, and division computations, respectively) during a 10-minute time period. At the end of the 10-minute math test, papers are collected and scored; the number of problems attempted and the number of problems correctly answered are generated as objective measures related to "academic productivity." A positive score indicates improvement.
Time Frame: Pre-dose to 10, 11, and 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number attempted
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Placebo
Number analyzed (Participants) | 159 | 157 | 157
Number attempted | 18.76 (3.065) | 28.03 (3.078) | -0.23 (3.073)

5. Secondary Outcome: Change From Pre-dose in the Permanent Product Measure of Performance of Measurement (PERMP) Math Test-Correctly Answered Score at 10, 11, and 12 Hours (Averaged) Post-dose
Description: as for outcome 4
Time Frame: Pre-dose to 10, 11, and 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number correct
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Placebo
Number analyzed (Participants) | 159 | 157 | 157
Number correct | 18.45 (2.461) | 28.02 (2.480) | -4.30 (2.474)

ADVERSE EVENTS:
Arm/Group | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/165 | 1/165 | 0/165
Other Adverse Events (participants affected / at risk) | 10/165 | 8/165 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg (N=165) | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg (N=165) | Placebo (N=165)
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dex-Methylphenidate Hydrochloride (Focalin XR) 30 mg (N=165) | Dex-Methylphenidate Hydrochloride (Focalin XR) 20 mg (N=165) | Placebo (N=165)
Decreased appetite (Metabolism and nutrition disorders) | 10 | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.